CLINICAL TRIAL: NCT06053242
Title: A Double-blinded, Randomized, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, and Effectiveness of CELZ-201-DDT Administered by Intramuscular Injection for the Treatment of Chronic Lower Back Pain in Patients With Degenerative Disc Disease
Brief Title: Safety, Tolerability, and Effectiveness of Intramuscular Injection of CELZ-201-DDT for the Treatment of Chronic Lower Back Pain
Acronym: ADAPT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Creative Medical Technology Holdings Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CELZ-201-ADAPT
Record Dates: First submitted 2023-09-17; First posted 2023-09-25 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low-back Pain; Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): Subjects in the low dose arm will receive a single administration of either 6x10^6 cells (n=8) or a placebo injection (n=2). Each subject will receive six paraspinal intramuscular injections (three injections per side) of either CELZ-201-DDT or placebo into the lumbar musculature under direct ultrasound guidance.
  Interventions: Drug: CELZ-201-DDT; Other: Placebo
- Medium Dose (Experimental): Subjects in the medium dose arm will receive a single administration of either 30x10^6 cells (n=8) or a placebo injection (n=2). Each subject will receive six paraspinal intramuscular injections (three injections per side) of either CELZ-201-DDT or placebo into the lumbar musculature under direct ultrasound guidance.
  Interventions: Drug: CELZ-201-DDT; Other: Placebo
- High Dose (Experimental): Subjects in the high dose arm will receive a single administration of either 60x10^6 cells (n=8) or a placebo injection (n=2). Each subject will receive six paraspinal intramuscular injections (three injections per side) of either CELZ-201-DDT or placebo into the lumbar musculature under direct ultrasound guidance.
  Interventions: Drug: CELZ-201-DDT; Other: Placebo

INTERVENTIONS:
Drug: CELZ-201-DDT — Subjects enrolled in the trial will receive CELZ-201-DDT at the specified dose into the lumbar paraspinal musculature. Each subject will receive a total of six injections, three injections on each side, under direct ultrasound guidance.
Other: Placebo — Subjects will receive a placbeo injection into the lumbar paraspinal musculature. Each subject will receive a total of six injections, three injections on each side, under direct ultrasound guidance.

SUMMARY:
The brief purpose of this research study is to learn about the safety, tolerability, and efficacy of paraspinal intramuscular injection of CELZ-201-DDT in patients with chronic lower back pain.

DETAILED DESCRIPTION:
This study is a double-blinded, randomized, placebo-controlled, dose escalation Phase 1/2a study. The objective is to determine the safety, tolerability, and efficacy of CELZ-201-DDT administered as an intramuscular injection for the treatment of lower back pain in patients with Degenerative Disc Disease. Subjects who meet all criteria for inclusion will be enrolled and randomized into either low, medium or high dose of CELZ-201-DDT versus Placebo, with a total of 30 subjects enrolled. Each dosing cohort will contain ten subjects (n=10), with eight subjects (n=8) receiving the investigational product and two subjects (n=2) randomized to receive placebo. Each subject will receive six paraspinal intramuscular injections (three injections per side) of either CELZ-201-DDT or placebo into the lumbar musculature under direct ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant to understand and the willingness to sign a written informed consent document.
* Between 18-80 years of age and may be of either gender or any race.
* Subjects must have failed at least two standard of care (SOC) therapies before being enrolled in the study: 1) exercise/physical therapy; 2) oral analgesic including nonsteroidal anti-inflammatory drugs (NSAIDs) and acetaminophen; 3) skeletal muscle relaxants. Subjects must have tried each SOC therapy for at least 3 months before failure is determined.
* Patients must have failed the SOC therapies within 12 months of enrollment in the clinical trial.
* Proof for one of the following tests already performed in the clinical care of the patient for lower back pain: 1) MRI scan demonstrating at least one disc level with grade II or greater disc degeneration using the Pfirrmann grading system; 2) Oswestry Disability Index for Back Pain score of 21-80%; 3) Visual Analogue Scale for pain of >5 on a scale of 0-10.
* Female subjects must not be breast feeding and must have no intention to become pregnant during the study, and she is using contraceptive drugs or devices.
* Any male subject must agree to use contraceptives and not donate sperm during the study.

Exclusion Criteria:

* History of cancer in the last five years.
* Spinal infections and spinal tumors.
* Renal insufficiency requiring dialysis or an eGFR of less than 60 mL/min/1.73m2.
* ALT, AST greater than 2 times or Total Bilirubin 1.5 times the upper limit of the normal range.
* Positive pregnancy test.
* History of blood cell diseases.
* Uncontrolled diabetes mellitus - HgA1c >8%.
* Uncontrolled hypertension defined as a systolic blood pressure of >140 mmHg or diastolic blood pressure of >90 mmHg at the time of screening. If subjects have their hypertension appropriately treated, then they would be eligible to enroll.
* Patients known to have any active infection, including infection of the injection site(s), and/or any active systemic or local infection.
* Patients on chronic immunosuppressive transplant therapy. Patients receiving <5 mg of Prednisone daily may be included.
* Subjects having a concomitant life-threatening disease in which their life expectancy is estimated to be less than 2 years.
* Recent smoking history or substance abuse (within six weeks).
* Heavy alcohol use (greater than 14 drinks per week for men or 7 drinks per week for women per NIAAA)
* Use of an investigational drug, device or product, or participation in a drug research study within a period of 30 days prior to receiving study treatment.
* Any patient who has received gene therapy in the past.
* Subjects who are currently on Schedule I or II controlled substances.
* Body Mass Index (BMI) > 40 kg/m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety of CELZ-201-DDT administered as intramuscular injections in subjects experiencing chronic lower back pain at a low, medium, or high dose. | 6 months
  The primary outcome will be evaluated by the incidence of grade 3 or 4 or serious adverse events in all dosing cohorts at 6 months.

SECONDARY OUTCOMES:
Evaluate the potential efficacy of CELZ-201-DDT therapy in terms of pain alleviation and improved mobility in subjects experiencing chronic low back pain. | 12 months
  The secondary outcome will be evaluated by change in pain as judged by the Visual Analogue Score (VAS), using a score of 0-10.
Evaluate the potential efficacy of CELZ-201-DDT therapy in terms of pain alleviation and improved mobility in subjects experiencing chronic low back pain. | 12 months
  The secondary outcome will be evaluated by change in disability as judged by the Oswestry Disability Index (ODI) for back pain.
Evaluate the potential efficacy of CELZ-201-DDT therapy in terms of pain alleviation and improved mobility in subjects experiencing chronic low back pain. | 12 months
  The secondary outcome will be evaluated by change in requirements for pain medications to manage back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Spine and Wellness Centers of America, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No